CLINICAL TRIAL: NCT03884855
Title: Randomised Controlled Trial to Evaluate the Benefit of Traditional Karate in Heart Failure During Cardiac Rehabilitation
Brief Title: Evaluation of the Benefit of Traditional Karate in Heart Failure for Cardiac Rehabilitation
Acronym: KAREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAREAD
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Cardiac Rehabilitation (Active Comparator): Patients benefit from a classic cardiac rehabilitation cycle during 3 months.
  Interventions: Other: Classical Cardiac Rehabilitation
- Karate Rehabilitation (Experimental): Patients benefit from cardiac rehabilitation cycle with traditional karate during 3 months.
  Interventions: Other: Karate rehabilitation

INTERVENTIONS:
Other: Classical Cardiac Rehabilitation — Patients benefit from classical cardiac rehabilitation during 3 months.
  Arms: Classical Cardiac Rehabilitation
Other: Karate rehabilitation — Patients benefit from cardiac rehabilitation with traditional karate during 3 months. Patients will have four 60-minute group sessions four times a week, during which they will have 45-minute individual exercises and 15-minute pairs of exercises. The course of the sessions has been protocolised.
  Arms: Karate Rehabilitation

SUMMARY:
Cardiac rehabilitation is based on physical activity which, usually, associates combination of a cycle ergometer or treadmill completed by gymnastics.

Some studies have been done with complementary physical activities such as tai chi or yoga integrated into the strategy of non-drug therapies. The tai chi study showed a tendency to improve the peak of VO2 in the tai chi group but which was not significant but also a significant improvement on secondary objectives such as quality of life, the increase in the 6-minute walk test and a decrease in the level of natriuretic peptides. A study of the effects of yoga after coronary artery bypass surgery showed at one year an improvement of the ejection fraction, the lipid profile and the state of anxiety of the patients. This study showed that the addition of yoga to conventional cardiac rehabilitation could improve cardiovascular risk factors especially in patients with abnormalities such as low HDL.

The physical activities offered in rehabilitation to improve physical performance are currently limited to cycling, treadmill or gymnastics. Many patients do not like cycling or treadmill, which limits their adherence to a cardiac rehabilitation program. Moreover, one of the main problems of rehabilitation is that after the rehabilitation cycle, a minority of patients continue the physical activity. Strategies for implementing home exercises have been tested to increase the level of physical activity after rehabilitation.

Cardiac rehabilitation has several components: correction of risk factors, optimization of treatment, physical activity to improve the physical abilities to exertion that are directly correlated to mortality.

Our hypothesis is that the implementation of a program of physical activity based on traditional karate would improve the physical abilities to effort and the quality of life of patients, to give a better psychological confidence to patients who, after a cardiovascular event such as acute coronary syndrome, bypass surgery or valvular surgery, have marked anxiety or depression. Rehabilitation, and especially physical activity, is one of the therapeutic means proposed. The interest of this study would be to be able to offer an additional activity for rehabilitation centers, to offer patients an activity in post-rehabilitation. In addition, interaction between patients could increase adherence to rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years
* Patient with heart failure
* Patient with impaired ejection fraction with Left ventricular ejection fraction ≤ 40%
* Patient affiliated with a health insurance plan
* Patient giving free, informed and express consent

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty
* Non-French speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
peak VO2 | Month 3
  The peak VO 2 will be measured during cardiac stress test at 3 month, at the end of cardiac rehabilitation.This peak VO2 measurement will be compared to peak VO2 at the Day 1, before cardiac rehabilitation.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | Day 1
  The following questions refer to patient's heart failure and how it may affect his life. This questionnaire quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | Month 3
  The following questions refer to patient's heart failure and how it may affect his life. The score will be compared to the responses to the questionnaire at Day 1. This questionnaire quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
DASS 21 scale | Day 1
  The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress. The scale will be completed at day 1. Each item is scored on a 4-point scale (0 = Did not apply to me at all, to 3 = Applied to me very much or most of the time). Sum the score of each item to get a total score. Higher scores indicate greater levels of distress.
DASS 21 scale | Month 3
  The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress. The scale will be completed at month 3, at the end of cardiac rehabilitation. Each item is scored on a 4-point scale (0 = Did not apply to me at all, to 3 = Applied to me very much or most of the time). Sum the score of each item to get a total score. Higher scores indicate greater levels of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DUC, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hôpital Corentin Celton, Issy-les-Moulineaux, Île-de-France Region